CLINICAL TRIAL: NCT04616105
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of REGN6490 in Healthy Japanese Volunteers
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetics of REGN6490 in Healthy Japanese Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R6490-HV-1993
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Single ascending subcutaneous (SC) dose 1 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- Cohort 2 (Experimental): Single ascending subcutaneous (SC) dose 2 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- Cohort 3 (Experimental): Single ascending subcutaneous (SC) dose 3 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo
- Cohort 4 (Experimental): Single ascending intravenous (IV) dose 4 of REGN6490 or matching placebo
  Interventions: Drug: REGN6490; Drug: Placebo

INTERVENTIONS:
Drug: REGN6490 — Single dose of REGN6490
Drug: Placebo — Placebo matching single dose of REGN6490

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of 3 single ascending subcutaneous (SC) doses and 1 single intravenous (IV) dose of REGN6490 in healthy first-generation Japanese adult participants

The secondary objectives of the study are:

* To characterize the pharmacokinetic (PK) profile of single SC and IV doses of REGN6490 in healthy first-generation Japanese adult participants
* Assess immunogenicity of REGN6490 in healthy first-generation Japanese adult participants dosed with a single IV or SC dose of REGN6490

ELIGIBILITY:
Key Inclusion Criteria:

1. Is a male or female first-generation Japanese participant 20 to 60 years of age (inclusive) at screening visit. First-generation Japanese subject must: (a) Be Japanese, born in Japan, and have both biologic parents and 4 biologic grandparents who are ethnically Japanese and born in Japan, (b) Have maintained a Japanese lifestyle, with no significant change since leaving Japan, including having access to Japanese food and adhering to a Japanese diet, (c) Have lived <10 years outside of Japan
2. Body mass index between 18 and 31 kg/m2 (inclusive) at screening visit
3. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and ECG's performed at screening and/or prior to administration of initial dose of study drug
4. Is in good health based on laboratory safety testing obtained at the screening visit
5. Willing and able to comply with clinic visits and study-related procedures
6. Provide informed consent signed by study participant

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, dermatological, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease, as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation
2. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
3. Has any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by study participation
4. Hospitalization (>24 hours) for any reason within 30 days of the screening visit
5. Is a current smoker, including e-cigarettes. Former smokers may be enrolled if they have stopped smoking for at least 3 months (90 days) prior to the screening visit

Note: Other protocol defined Inclusion/Exclusion criteria apply

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | Up to Week 16
  TEAEs include abnormal laboratory testing, vital signs and electrocardiograms (ECGs)

SECONDARY OUTCOMES:
Serum Concentration of REGN6490 over time | Up to Week 16
Incidence of Treatment-Emergent REGN6490 Anti-Drug Antibodies (ADAs) | Up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/